CLINICAL TRIAL: NCT01293812
Title: A Randomized Double-blind Trial Comparing the Effect on Pain of an Oral Sucrose Solution Versus Placebo in Children 1 to 3 Months Old Needing Venipuncture
Brief Title: Effect on Pain of Oral Sucrose Versus Placebo in Children 1 to 3 Months Old Needing Venipuncture
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: Canadian Association of Emergency Physicians (Industry)
Responsible Party: Principal Investigator, Serge Gouin, Asociate Professor, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Sucrose#3236
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sucrose po (Experimental): 88% sucrose solution (Syrup B.P.). The pharmacy will provide 2 syringes labeled "sucrose study" calculated to provide a 2 ml dose of a 88% sucrose solution.
  Interventions: Drug: 88% sucrose po solution
- placebo po (Placebo Comparator): The pharmacy will provide 2 syringes labeled "sucrose study" calculated to provide a 2 ml dose of a color, consistency- and odor-matched placebo to the sucrose solution in identical packagings (2 syringes per patient in the case the dose needs to be repeated).
  Interventions: Drug: placebo po

INTERVENTIONS:
Drug: 88% sucrose po solution — 88% sucrose solution (Syrup B.P.) The pharmacy will provide 2 syringes labeled "sucrose study" calculated to provide a 2 ml dose of a 88% sucrose solution or a color, consistency- and odor-matched placebo in identical packagings (2 syringes per patient in the case the dose needs to be repeated).
  Arms: sucrose po
Drug: placebo po — The pharmacy will provide 2 syringes labeled "sucrose study" calculated to provide a 2 ml dose of a solution or a color, consistency- and odor-matched placebo to the sucrose solution in identical packagings (2 syringes per patient in the case the dose needs to be repeated).
  Arms: placebo po

SUMMARY:
Background : Previous studies suggest that early recognition and treatment of pain among children is important for their cognitive development and their future response to pain throughout their life. Oral sweet solutions have been accepted as effective pain reducing agents for procedures in the neonatal population. To date, there have been a limited number of published clinical trials in an emergency setting studying this type of intervention among infants and these studies have shown conflicting results.

Objective : To compare the efficacy of an oral sucrose solution versus placebo in reducing pain in children 1 to 3 months of age during venipuncture in the Emergency Department (ED).

Methods : A single-center, randomized, double-blind, placebo controlled clinical trial will be conducted in an urban tertiary care pediatric university-affiliated hospital ED. The study population is all infants from 1 to 3 months of age requiring venipuncture as part of their planned ED management. Study participants will be randomly allocated to receive 2 ml of a 88% sucrose solution or 2 ml of a placebo solution. The primary outcome measure is the difference in pain levels during the venipuncture in the study population as assessed by the Face, Legs, Activity, Cry and Consolability Pain Scale (FLACC). Secondary outcome measures will evaluate differences of pain levels using the Neonatal Infant Pain Scale (NIPS). Crying time and changes in heart rate during the procedure will be recorded. Side effects and adverse events will also be noted. The investigators will also measure the number of successful venipunctures at the first attempt. Based on previously reported data, using an alpha value of 0,05, a power of 90% and using a 2-point difference in mean FLACC scores as clinically significant difference, approximately 41 patients per group will be needed considering a drop-off value of 25%. Patients' characteristics and outcomes will be compared using the Pearson Chi-square test for categorical variables and the Student's T test for continuous variables. A intention to treat analysis will be performed.

DETAILED DESCRIPTION:
INTRODUCTION AND JUSTIFICATION

Acute pain is one of the most common adverse stimuli experienced by children, occurring as a result of injury, illness, and necessary medical procedures[1]. The American Academy of Pediatrics (AAP) and the American Pain Society (APS) have jointly issued a statement promoting the responsibility of paediatricians as leaders and advocates to ensure the humane and competent treatment of pain and suffering in all infants, children, and adolescents[1]. In Emergency Departments (ED), children undergo many painful procedures, such as bladder catheterization, capillary blood tests, venipuncture and lumbar puncture. All these procedures are associated with increased anxiety, avoidance, somatic symptoms, and increased parental distress[1]. Numerous myths, insufficient knowledge among caregivers, and inadequate application of knowledge contribute to a lack of effective pain management among infants[1].

Long-term effects of unmanaged pain in human infants have been shown to include permanent impairment of elements of cognitive development, such as learning, memory, and behaviour[2], and increased somatisation in childhood[3]. The plasticity of the developing brain and the changes that occur in response to painful stimuli[4] also contribute to altered perceptions of pain later in life[5-6]. Early painful experiences affect children's future responses to analgesia. Weisman et al[7] found that inadequate analgesia in young children during procedures diminished the effects of adequate analgesia during subsequent procedures. Many studies have suggested that the prompt and accurate recognition and treatment of pain in young infants is important for their immediate comfort and for their best possible lifelong development[8]. Despite the recent interest in paediatric pain assessment, prevention and treatment, many children do not receive adequate management to alleviate pain[1, 8-9]. The ideal pre-procedural analgesic for minor invasive procedures would be a cost-effective, inexpensive, short-acting agent with few associated risks[10].

The use of sucrose has been well studied for certain procedures in the patients of the neonatal intensive care unit and in the newborn nursery settings, particularly for venous blood draws, capillary blood tests and circumcision[11-13]. In these studies[11-13], infants receiving oral sucrose solutions before procedures cried less and had overall decreased behavioural pain responses when compared with those receiving placebo. Furthermore, sucrose has been shown to be a safe intervention with no serious life-threatening adverse events and only few reported side effects consisting of minimal coughing with administration[14]. Sucrose is inexpensive, short acting, non-sedating, easily administered and non-invasive. Administration of sucrose does not require additional training and does not expose the infant to risks greater than those associated with breast or bottle feeding.

Summaries of randomized controlled trials among hospitalized neonates of 32 to 40 weeks of gestation suggest that a single dose of 0,5 to 2 mL of 12% to 50% sucrose delivered by non-nutritive sucking via a pacifier for 2 minutes before a painful event is safe[15] and effective in decreasing physiologic (heart rate, respiratory rate and oxygen saturation)[16-17]. It is also effective in minimizing behavioural pain indicators (crying, facial expression and motor activity)[16, 18] and in reducing overall composite pain scale scores[16]. A Cochrane systematic review concluded that sucrose is safe and effective in reducing procedural pain from single short procedural events in neonates, but an optimal dose could not be identified due to inconsistency in effective sucrose dosage among studies[19]. A review of published studies reported that sucrose or glucose in healthy term or preterm infants during single episodes of heel lancing, venipuncture or intramuscular injection is effective[20]. However, uncertainties remain beyond the neonatal period, given the limited number of published studies [20].

A growing number of studies looking at infants undergoing immunizations suggest that this analgesic effect may extend past the neonatal period and into infancy[21-26]. Nevertheless, the upper limit of this effect is unknown in terms of age and appropriate sucrose dosage. Two studies have examined the effectiveness of sweet solutions as an analgesic in the paediatric ED. A randomized controlled trial in an emergency setting of sucrose and/or pacifier for infants receiving venipuncture conducted by Curtis and al[27] among infants of 0 to 6 months demonstrated a trend in reducing pain among the sub-group of infants of 0 to 3 months. However, this study showed no difference in pain scales after 3 months of age. Also, in a study examining the effect of sucrose during bladder catheterization, the subgroup of infants 1 to 30 days old who received a sweet solution showed smaller changes in pain scores, were less likely to cry during catheterization and returned to baseline more quickly, in comparison with the placebo group[14]. However, among children of 31 to 90 days, there was no statistically significant difference.[14].

Also, studies have used varieties of concentrations of sucrose (e.g. Rogers had used sucrose 24%[14], Curtis had used sucrose 44%[27] and Lewindon had used sucrose 75%[24]). Systematic reviews of the current literature have been unable to demonstrate superiority of one concentration of a sweet solution over another[28], but many studies suggest that higher concentrations of sweet solutions seem more effective[25, 29-32]. Therefore, the investigators chose to study the effect of a sweet solution named syrup B.P. (product by Laboratoire Atlas inc.) which contains 88% of sucrose. This solution is already commonly used in the population of infants up to 3 months of age and it is safe (e.g. prednisone syrup or codeine syrup are made using this syrup). A 2 ml dose of 88% sucrose contains the same amount of carbohydrates as 25 ml of infant milk formulas which contain approximately 7,5g/100 ml[33]. Also, 88% sucrose has the same concentration of sugar as many other medications which are commonly used in infants, such as oral antibiotics, oral steroid solutions and other pain medications (e.g. codeine syrup). This syrup is of particular interest as it is of low cost ($9,58 for a bottle of 2000 ml), universally available, stable and viable for approximately three months. Therefore, the procedure studied here would be easy to apply in most clinical settings.

Finally, the painful procedure chosen for our study is venipuncture (indwelling catheter with or without drawing of blood samples). Venipunctures are frequently performed in the ED in this age group. In fact, in our study center, the CHU Ste-Justine, approximately 15 patients of 1 to 3 months require venipuncture as a part of their investigation each month.

To date, there are no pain scales which have been validated precisely for the age group studied in our project. However, the Face, Legs, Activity, Cry and Consolability (FLACC) scale is recommended by the IMMPACT group (Initiative on Methods, Measurement and Pain Assessment in Clinical Trials)[34]. FLACC is an easily applicable pain scale in which the observer scores a patient for 5 categories, from 0 to 2 points, for a total score of maximum 10 points (Table 1). The validity and reliability of this pain scale has been established in the past for children from 2 months to 7 years[35]. Validity was evaluated by comparing the FLACC scale with the Objective Pain Scale and demonstrated that both tools showed similar behaviours (r=0.80; p<0.001)[35]. The interrater reliability between 2 observers was considered good (r[87]=0.94; p<0.001) with a kappa value greater than 0,50 for each category[35]. Therefore, this pain scale was chosen as the measure of our primary outcome, in our population of infants from 1 to 3 months old. Furthermore, the Neonatal Infant Pain Scale (NIPS)[36] (Table 2) is a well validated pain scale for newborns up to 1 month of age[37]. This pain scale was chosen as a secondary outcome. The investigators hypothesize that using one pain scale validated in infants up to 1 month of age and another validated in infants older than 2 months of age will allow us to assess pain in infants from 1 to 3 months of age best, given current available tools. Furthermore, several other patient parameters will be used to corroborate findings.

HYPOTHESIS The investigators believe that providing an oral sucrose solution during venipuncture will decrease pain levels in infants 1 to 3 months of age.

OBJECTIVES Our primary objective is to compare the efficacy an oral 88% sucrose solution to a placebo solution in reducing pain as assessed by the Face, Legs, Activity, Cry and Consolability scale in children of 1 to 3 months during venipuncture in the Emergency Department (ED). Our secondary objectives are to asses changes in pain levels as per the NIPS scores. The investigators will also measure variations of heart rate and crying time. Any side effects will also be reported. The investigators will also measure the number of successful venipunctures at the first attempt.

ELIGIBILITY:
Inclusion Criteria:

* Infants from 1 to 3 months (one month or more but less than 3 months old) of actual age (not corrected) requiring a venipuncture as a part of their planned ED management during weekdays from 9h to 17h.

Exclusion Criteria:

1. Preterm infants (i.e. born < 37 weeks)
2. Acute respiratory illness
3. Chronic cardio-pulmonary condition
4. Assisted ventilation (such as tracheostomy or oxygen dependance)
5. Technology dependant (such as enteral feeding tube)
6. Developmental delay
7. Oropharyngeal malformation or dysfunction (such as cleft palate or micrognathia)
8. Metabolic disease
9. Previous participation in this study
10. Painful procedures in the preceding 60 minutes (bladder catheterization, vesical puncture, lumbar puncture, capillary blood tests)
11. Parental language barrier (French and/or English)

Ages: 1 Month to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2011-02; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Difference in pain scores related to venipuncture in the study population as assessed by the Face, Legs, Activity, Cry and Consolability Pain Scale before the administration of sucrose and one minute after the venipuncture | one minute

SECONDARY OUTCOMES:
The difference in pain scores using the Neonatal Infant Pain Scale (NIPS). | one minute

CONTACTS AND LOCATIONS:
Overall Officials: Serge Gouin, MDCM, FRCPC, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Ste-Justine, Montreal, Quebec, Canada